CLINICAL TRIAL: NCT06040671
Title: Objective Evaluation of the Effect of Oculoplastic Operations Using the Vectra M 3D Imaging System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 28/RVO-FNOs/2021
Record Dates: First submitted 2022-10-31; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Eyelid Ptoses; Ectropion Eyelids; Entropion;Eye
Keywords: Vectra M3 device; Eyelid Ptoses; stereo photographic system; eyelid surgery
MeSH Terms: conditions — Blepharoptosis; Ectropion; Entropion

STUDY DESIGN:
Intervention Model Description: The study subjects will be divided into two groups.
Masking Description: No masking is used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral canthal hinge surgery patients (Experimental): Patients undergoing lateral canthal hinge surgery will be enrolled in this group.
  Interventions: Other: Vectra M3 imaging
- Ptosis surgery patients (Experimental): Patients undergoing ptosis surgery will be enrolled in this group.
  Interventions: Other: Vectra M3 imaging

INTERVENTIONS:
Other: Vectra M3 imaging — Study subjects from both arms will undergo Vectra M3 imaging to evaluate the result of the surgery.

SUMMARY:
An objective assessment of that part of the spectrum of ophthalmic eyelid surgeries that focuses on correcting the position of entropy (e.g. ectropion, ptosis surgery) is very difficult - although it is possible to use different measuring parameters (distance of pupillary reflexes from the edges of the eyelid), comparing different distances on the face, exophthalmometry or the lid laxity test - the so-called snap-back test, but all these methods are based either on the subjective assessment of the examiner or on the correctness of the attached ruler, and their objectivity is therefore very low.

DETAILED DESCRIPTION:
The goal of the project is to develop a methodology for evaluating the results of operations using a stereo photographic system, to objectively evaluate the functionality and results of various eyelid operations, and subsequently to expand the use of the device in other ophthalmological indications.

Different files will be created where the effect of different operations will be monitored in parallel.

Lateral canthal hinge surgery will be evaluated in the pilot group, and ptosis surgery through an anterior approach will be evaluated in the second group.

In all patients, the position of the eyelids, their change before and after surgery, the periorbital volume, and the relation of the eyelids to the periorbital landscape will be assessed metrically.

The Vectra M3 device will be used for the measurement.

The expected cohort size is 40 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* Eyelid ptosis
* Eyelid entropion
* Eyelid ectropion

Exclusion Criteria:

* Refusal to participate in the study
* Not signing the Informed Consent Form
* Inability/reluctance to cooperate in the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Distance between anatomical points on the face | 6 months
  In all patients, distance between 52 anatomical-topographical points on the face will be measured in millimetres (mm) - change of the position of the eyelids before and after surgery (distance in mm), the relation of the eyelids to the periorbital landscape (distance in mm)
Periorbital volume measurement | 6 months
  In all patients, the periorbital volume (volume in mm3) will be assessed metrically.

SECONDARY OUTCOMES:
The possibility to use the Vectra M 3D Imaging System in other ophthalmological indications | 3 years
  The suitability (YES/NO) of using the Vectra M 3D Imaging System in other ophthalmological indications will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kopecký, MD,PhD,FEBO, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers; however, the data may be provided upon request.